CLINICAL TRIAL: NCT06652633
Title: A Long-term Follow-up Study for Patients Treated With Galapagos CAR T-cell Therapies
Brief Title: Long-term Follow-up of Participants Treated With Galapagos Chimeric Antigen Receptor (CAR) T-cell Therapies
Acronym: Hesperia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LTF-CL-001; 2023-510173-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hematological Malignancies
Keywords: CAR T-cell therapy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Previously treated participants with GLPG CAR T-cell therapy (Experimental): All participants who have been treated with a Galapagos CAR T-cell therapy
  Interventions: Genetic: GLPG CAR T-cell therapy

INTERVENTIONS:
Genetic: GLPG CAR T-cell therapy — No investigational products will be administered to participants in this study.

SUMMARY:
This is a long-term follow-up study for participants treated with Galapagos (GLPG) CAR T-cell therapies to evaluate the long-term safety and efficacy of GLPG CAR T-cell products for 15 years post infusion.

Per Health Authorities guidelines for gene therapy medicinal products that utilize integrating vectors (e.g. lentiviral vectors), long term safety and efficacy follow up of treated patients is required. The purpose of this study is to monitor all participants exposed to GLPG CAR T-cell therapies for 15 years following their last CAR T-cell infusion to assess the risk of delayed adverse events (AEs) and the long-term benefit/risk profile and to monitor for replication-competent lentivirus (RCL) and CAR-T cell persistence.

ELIGIBILITY:
Inclusion Criteria:

* All participants who have been treated with a Galapagos CAR T-cell therapy in a clinical trial or Managed Access Program.

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2039-07 (Estimated); Study Completion 2039-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with targeted adverse events (AEs) | From infusion up to 15 years
Percentage of participants with detectable CAR transgene levels in peripheral blood | From infusion up to 15 years
Percentage of participants with serious AEs (SAEs) considered related to the Galapagos CAR T-cell therapy | From infusion up to 15 years
Percentage of participants with at least 1% of T-cells in the blood sample or positive new malignancies | From infusion up to 15 years
Percentage of participants with detectable replication-competent lentivirus (RCL) in peripheral blood | From infusion up to 15 years
Percentage of participants who died with causes | From infusion up to 15 years

SECONDARY OUTCOMES:
Percentage of participants with disease progression | From infusion up to 15 years
Time to subsequent anticancer therapy | From infusion up to 15 years
Overall survival | From infusion up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (6):
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - Centre Hospitalier Universitaire (CHU) De Liège, Liège
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Leids University Medical Center (LUMC), Leiden
- Hospital Clinic De Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No